CLINICAL TRIAL: NCT03927807
Title: A Comparison of the Efficacy and Safety of Repetitive Hourly Dose of Oral Misoprostol and Two Hourly Dose Oral Regimens for Cervical Ripening and Labor Induction
Brief Title: Oral Misoprostol Solution in Labor Induction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esam salah mohamed hagag, Director,clinical research, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: misoprostol in induction
Record Dates: First submitted 2019-04-20; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Labour,Induced
Keywords: misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repetitive hourly dose of oral misoprostol (Experimental): The dose will be 10 microgram oral misoprostol that will be administered hourly up to 12 doses or till onset of regular uterine activity.
  Interventions: Drug: Misoprostol
- two hourly dose of oral misoprostol (Experimental): The dose will be 20 microgram oral misoprostol solution that will be administered every 2 hours up to 6 doses or till onset of regular uterine activity.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — This study will include 150 pregnant women who fulfill the inclusion criteria and will be subdivided in two groups.
  Group1 will receive repetitive hourly dose of oral misoprostol solution equal to 10 microgram up to 12 doses or regular uterine activity.
  Group2 will receive oral misoprostol solution every two hours as 20 microgram up to 6 doses or regular uterine activity.

SUMMARY:
This study compares safety and efficacy between repetitive hourly dose of oral misoprostol and two hourly dose oral regimens for cervical ripening and labor induction.

DETAILED DESCRIPTION:
Misoprostol is an effective agent for the induction of labor.existing guidelines recommend oral misoprostol solution every two hours.However,more research is required to optimize the use of oral misoprostol solution for labor induction.The current study is to compare efficacy and safety of repetitive hourly dose of oral misoprostol solution with two hourly dose of oral misoprostol solution for cervical ripening and labor induction.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparas
* Term pregnancy(equal or more than 37 wks)
* Bishop score <6
* Cephalic presentation
* reassuring fetal heart rate pattern
* Not in labor ( no uterine contractions)
* Clinically adequate pelvis
* Singleton live pregnancy

Exclusion Criteria:

* Allergic to misoprostol or prostaglandin analogues
* Previous uterine scar( cesarean section,hysterotomy,myomectomy)
* Multiple fetal gestations
* Fetal demise
* Preterm labor
* Malpresentations
* Non reactive cardiotocography at admission
* Cephalo pelvic disproportion
* Fetal macrosomia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — 150 pregnant women who fulfill inclusion criteria.these will be subjected to history taking,physical examination,counseling and signing a written consent will be taken from each case.
Enrollment: 150 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-18 (Estimated); Study Completion 2020-01-18 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | 24 hours from the first dose of induction till delivery
  Successful vaginal delivery within 24 hours from starting induction of labor or cesarean section delivery after failed trial of induction.

SECONDARY OUTCOMES:
Adverse maternal outcomes | in 24 hours
  As uterine hyper stimulation,fever,vomiting,shivering,nausea
Adverse neonatal outcomes | 24 hours post partum
  As neonatal intensive care unit admission,non reassuring fetal heart rate

CONTACTS AND LOCATIONS:
Overall Officials: essam sa hagag, MBBCh, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel.requestors will be required to sign a data access agreement.
URL: http://bethesda.org

REFERENCES:
- [Result] 27986461